CLINICAL TRIAL: NCT00348530
Title: Prospective, Randomized Comparison of Therapy With Verapamil or Carvedilol on Long-Term Outcomes of Patients With Chronic Heart Failure Secondary to Non-Ischemic Cardiomyopathy
Brief Title: Carvedilol Versus Verapamil in Chronic Heart Failure Secondary to Non-Ischemic Cardiomyopathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Silesia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CavsBe.2006
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2006-10-18 (Estimated); Status verified 2006-01

CONDITIONS: Systolic Heart Failure; Myocardial Disease; Cardiomyopathy
Keywords: Systolic heart failure; Therapy; Cardiomyopathy
MeSH Terms: conditions — Heart Failure, Systolic; Cardiomyopathies | interventions — Verapamil

INTERVENTIONS:
Drug: Verapamil

SUMMARY:
Accumulated clinical and experimental data suggest that dysfunctional coronary microcirculation plays a pivotal role in the progression of heart failure despite an optimal therapy used. Therefore, we hypothesize that improvement in microvascular function by calcium antagonist, verapamil may result in additional clinical benefit. Thus, the aim of this study is to compare the effect of treatment with verapamil or carvedilol on long-term outcomes in stable, chronic heart failure secondary to non-ischemic cardiomyopathy.

DETAILED DESCRIPTION:
Heart failure, irrespective of its etiology may be viewed as a progressive disorder initiated by a different events and sustained by a multifaceted pathophysiological mechanisms. Regardless of the nature of the initiating events and optimized therapy used, loss of functioning cardiac myocytes developed and the disease progressed. One potential explanation for such progression is that not all pathological mechanisms underlying the disease are antagonized enough by currently used therapeutic strategy. Accordingly, impaired myocardial perfusion secondary to microvascular dysfunction has been postulated to play a major role in the progression of heart failure despite standard therapy for heart failure (1). It has been hypothesized that diffuse subendocardial ischemia due to altered coronary physiology may contribute to the global cardiac dysfunction seen in heart failure patients (2). Accordingly, coronary endothelial dysfunction at the microvascular and epicardial level in patients with acute-onset idiopathic dilated cardiomyopathy and chronic congestive heart failure has been reported (3,4) Thus, taking all mentioned above into account, the improvement in endothelial function and diminishing of subendocardial ischemia with calcium antagonists may be promising in terms of using these drugs for therapy of patients with stable chronic heart failure. The previous randomized study (5) and our long-term pilot study support this point of view.

1. Neglia D, Michelassi C, Trivieri MG, et al. Prognostic role of myocardial blood flow impairment in idiopathic left ventricular dysfunction. Circulation 2002;105:186-193.
2. Unverferth DV, Magorien RD, Lewis RP, et al. The role of subendocardial ischemia in perpetuating myocardial failure in patients with nonischemic congestive cardiomyopathy. Am Heart J 1983;105:176-179.
3. Mathier MA, Rose GA, Fifer MA, et al. Coronary endothelial dysfunction in patients with acute-onset idiopathic dilated cardiomyopathy. J Am Coll Cardiol 1998;32:216-224.
4. Chong AY, Blann AD, Patel J, et al. Endothelial dysfunction and damage in congestive heart failure. Relation of flow-mediated dilation to circulating endothelial cells, plasma indexes of endothelial damage, and brain natriuretic peptide. Circulation 2004;110:1794-1798.
5. Figulla HR, Gietzen F, Zeymer U, et al. Diltiazem improves cardiac function and exercise capacity in patients with idiopathic dilated cardiomyopathy. Results of diltiazem in dilated cardiomyopathy trial. Circulation 1996;94:346-352.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure (NYHA II and III; LV ejection fraction, ≤ 35%) secondary to non-ischemic cardiomyopathy. Stable condition at least 6 months before enrollment on conventional therapy (beta-blockers, ACE inhibitors and diuretics).

Exclusion Criteria:

* improvement in clinical status on conventional therapy in out-patients period preceded hospitalization
* any changes narrowing epicardial coronary arteries in coronary angiography,
* insulin dependent diabetes,
* valvular heart disease (except the relative mitral regurgitation),
* endocrine disease,
* lack of written informed consent,
* significant renal and liver diseases,
* drug or alcohol abuse,
* therapy with steroids or calcium blockers within 3 months before screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2006-01; Study Completion 2007-12

PRIMARY OUTCOMES:
NT-proBNP; LVEF(radionuclide ventriculography; LVFS; LVDD/LVSD, NYHA class, V02, 6 min walking test, MLWHFQ.

SECONDARY OUTCOMES:
Death; Heart transplantation; Readmission to hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Romuald Wojnicz, MD, PhD, Principal Investigator — Medical University of Silesia
Locations (1):
- Silesian Center for Heart Disease, IIIrd Department of Cardiology, Silesian Medical University, Zabrze, Poland